CLINICAL TRIAL: NCT00420823
Title: A 12-week, Parallel, Double-blind, Randomised, Placebo-controlled Adjunctive Study of Taurine 4 Grams in 128 Patients With First-episode Psychosis Receiving Antipsychotic Treatment.
Brief Title: A Study of Taurine in Patients With First-episode Psychosis Receiving Antipsychotic Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Stanley Medical Research Institute (Other); Southern Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHREC 2006/040; SMRI Grant ID Number 06T-811 (Other Grant/Funding Number: Stanley Medical Resarch Institute)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Psychotic Disorders
Keywords: First Episode Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo pill (Placebo Comparator): 4 placebo pills daily for 3 months
  Interventions: Drug: Taurine 4g
- Taurine 4g (Experimental): Taurine 4g daily comprising four 1g pills
  Interventions: Drug: Taurine 4g

INTERVENTIONS:
Drug: Taurine 4g

SUMMARY:
The purpose of this study is to determine whether Taurine 4g is effective with antipsychotic medication in the treatment of First Episode Psychosis.Taurine may have an effect on cognition and symptoms. We are examining changes in symptoms and cognition over a 3 month period.

DETAILED DESCRIPTION:
The core rationale of this study will be to prospectively investigate whether Taurine will improve and /or protect cognitive functioning and improve symptomatology in a cohort of 128 first episode psychosis patients.This is a randomized, double blind placebo controlled add on standard therapy trial of Taurine 4g , in young patients between 18-25 presenting to ORYGEN Youth Health a sub program of Melbourne Health and RAPPS, a subprogram of Southern Health with a first psychotic episode . Taurine will be compared with placebo added to standard treatment for a period of 12 weeks in a double blind fashion.Primary outcome measures will be psychopathology and cognition (MATRICS.

Secondary outcome measures will be tolerability and safety measures (drop-out rates, general side effect scale (UKU).

Patients who give informed consent will be randomised to receive treatment with Taurine 4g daily or placebo for 12 weeks.

Patients will be randomised by a dynamic randomisation method called minimization which allocates patients to treatment group by checking the allocation of similar patients already randomised, and allocating the next treatment group "live" to best balance the treatment groups across all stratification variables. The minimization will be carried out by the NHMRC clinical trials centre in Sydney , and the patient will be randomized to either placebo or vitamin.

Each patient will collect their tablets from the clinical trials pharmacy. The Clinical Trials Pharmacy will dispense either vitamin or placebo. All study personnel and participants will be blinded to treatment assignment for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* Between 18 and 25 years of age
* First Episode Psychosis
* Attending ORYGEN Youth Health, a geographical based catchment area service for young people aged between 15 and 25.

Exclusion Criteria:

* Organic disorders presenting with a psychotic syndrome (e.g. brain tumour, temporal lobe epilepsy, HIV encephalopathy)
* Mental retardation (unable and/or unlikely to give appropriate information of symptomatology or side-effects (IQ approximately lower than 80)
* History of clinically significant physical illness (e.g. terminal cancer, renal dialysis)
* History of brain surgery
* History of brain infarction
* Pregnant or lactating women or women of childbearing potential not using an acceptable method of contraception.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognition (MATRICS Composite score) at 3 months
Symptomatology at 3 months

SECONDARY OUTCOMES:
Safety at 3 months
Tolerability at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Colin P O'Donnell, MB,MRCPsych, Principal Investigator — ORYGEN Research Centre , ORYGEN Youth Health,Department of Psychiatry,
Locations (2):
- Australia (2):
  - ORYGEN Youth Health, Melbourne, Victoria
  - RAPPS programme, Southern Health, Melbourne, Victoria

REFERENCES:
- [Derived] O'Donnell CP, Allott KA, Murphy BP, Yuen HP, Proffitt TM, Papas A, Moral J, Pham T, O'Regan MK, Phassouliotis C, Simpson R, McGorry PD. Adjunctive Taurine in First-Episode Psychosis: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study. J Clin Psychiatry. 2016 Dec;77(12):e1610-e1617. doi: 10.4088/JCP.15m10185. PMID 27835719